CLINICAL TRIAL: NCT03054285
Title: Does Short-Term Anti-Seizure Prophylaxis After Traumatic Brain Injury Decrease Seizure Rates?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Richard Gonzalez, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209136
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Seizures; Traumatic Brain Injury
Keywords: Seizures; Traumatic Brain Injury; Prophylaxis; Levetiracetam
MeSH Terms: conditions — Seizures; Brain Injuries, Traumatic | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: The intervention study model is a randomized block design using a 1:1 allocation scheme
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- No seizure prophylaxis (No Intervention): Participants randomized to this arm will not receive anti-seizure prophylaxis
- Seizure Prophylaxis (Experimental): Participants randomized to this arm will receive the anti-seizure prophylaxis drug Levetiracetam for seven days post traumatic brain injury.
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — Participants assigned to the experimental arm will receive a seven day course of levetiracetam for post-traumatic brain injury
  Other Names: Keppra
  Arms: Seizure Prophylaxis

SUMMARY:
The primary objective of this study is to prospectively assess in randomized fashion whether short term anti-seizure prophylaxis in traumatic brain injured patients decreases the incidence of seizures in the early post-injury period. A secondary objective is to evaluate whether there are differences in mortality, hospital length of stay, functional outcome at hospital discharge, hospital cost, discharge status (home, rehabilitation facility, etc.) for patients who receive and do not receive anti-seizure prophylaxis.

DETAILED DESCRIPTION:
The efficacy of anti-seizure prophylaxis in head injury patients remains controversial. Current recommendations for the use of anti-seizure prophylaxis are based upon a single institution study that has not been reproduced with other studies contradicting their conclusions. The proposed study will be a randomized prospective study at Loyola University Medical Center to assess the efficacy of anti-seizure prophylaxis in patients who have suffered traumatic brain injury (TBI). Patients with suspected TBI will undergo computed tomographic (CT) scan of the head. Following identification of TBI on CT scan, patients will be randomized to one of two study groups. Patients will be randomized to receive a seven-day course of anti-seizure prophylaxis with levetiracetam (UCB Pharma Inc.; Keppra) or randomized to a study group that will not receive anti-seizure prophylaxis. Patients will be consented prior to entry in the study. Patients will be followed for a total of seven days post injury for clinical signs of seizure activity. Additionally, patients will be assessed at one month post injury for clinical signs of seizure activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have suffered intracranial injury identified by CT Scan

Exclusion Criteria:

* Age less than 18
* Pregnant patients
* Death in ED
* Seizure history or use of antiepileptic medication prior to admission
* Contraindication to study drug
* Any post-injury seizures prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Seizures (count of seizures) | 30 days
  For all patients, the count of seizures will be recorded and compared between the two arms

SECONDARY OUTCOMES:
Mortality | 30 days
  For all patients, days from head injury to death or last follow-up will be recorded and compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gonzalez, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Pitkanen A, Immonen R. Epilepsy related to traumatic brain injury. Neurotherapeutics. 2014 Apr;11(2):286-96. doi: 10.1007/s13311-014-0260-7. PMID 24554454
- [Background] Torbic H, Forni AA, Anger KE, Degrado JR, Greenwood BC. Antiepileptics for seizure prophylaxis after traumatic brain injury. Am J Health Syst Pharm. 2013 Dec 1;70(23):2064, 2067. doi: 10.2146/ajhp130439. No abstract available. PMID 24249751
- [Background] Cranley MR, Craner M, McGilloway E. Antiepileptic prophylaxis following severe traumatic brain injury within a military cohort. J R Army Med Corps. 2016 Apr;162(2):109-14. doi: 10.1136/jramc-2014-000392. Epub 2015 Feb 24. PMID 25712562
- [Background] Temkin NR, Dikmen SS, Wilensky AJ, Keihm J, Chabal S, Winn HR. A randomized, double-blind study of phenytoin for the prevention of post-traumatic seizures. N Engl J Med. 1990 Aug 23;323(8):497-502. doi: 10.1056/NEJM199008233230801. PMID 2115976
- [Background] Young B, Rapp RP, Norton JA, Haack D, Walsh JW. Failure of prophylactically administered phenytoin to prevent post-traumatic seizures in children. Childs Brain. 1983;10(3):185-92. doi: 10.1159/000120113. PMID 6409521
- [Background] Bhullar IS, Johnson D, Paul JP, Kerwin AJ, Tepas JJ 3rd, Frykberg ER. More harm than good: antiseizure prophylaxis after traumatic brain injury does not decrease seizure rates but may inhibit functional recovery. J Trauma Acute Care Surg. 2014 Jan;76(1):54-60; discussion 60-1. doi: 10.1097/TA.0b013e3182aafd15. PMID 24368357